CLINICAL TRIAL: NCT03325478
Title: Qualitative Assessment of the French Brief Contact Intervention "Stay in Contact" in Suicide Prevention
Brief Title: Qualitative Assessment of the Brief Contact Intervention "Stay in Contact" in Suicide Prevention
Acronym: EVAREST2
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01023-50
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-08

CONDITIONS: Suicide and Self-harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Over the phone interviews on the BCI "Stay in Contact" — This study used phone call interviews on a BCI "Stay in Contact", 6 months after suicide attempt behavior.The questionnaire used for the interview of included suicide attempters was pilot tested to assess acceptability and feasibility of the study. It included 24 questions, which were based on literature's data.They covered seeking care and help items and assess the subjective quality appreciation of medical care in the PED and on the BCI.Closed-ended and multiple-choice questions were mixed. Included patients were informed that the questionnaire was anonymous and that seeking their views and feedbacks would help adjusting the implementation of follow-up interventions closer to their needs.The baseline interviews were conducted on the phone, on weekdays, during a mean time of 10 to 15minutes by a trained resident in psychiatry as the only interviewer.

SUMMARY:
Background: For 40 years, brief contact interventions (BCIs) have been presented as promising approaches in suicide prevention but patient's experiences of BCIs are less investigated.

Aim: Understand mechanisms of BCIs after suicide attempt, through patient's experience of a French BCI "Stay in contact" and assess its impact on seeking care during suicidal crisis.

Method:This is a single-center, non-interventional, prospective qualitative study using phone call interview on a BCI, 6 months after suicide attempt behavior.

Statistical analysis

Data were analyzed using statistical software (Version 9.4, SAS Institute Inc., Cary, North Carolina, USA). Chi-squared test was used to assess qualitative variables and t-test to evaluate quantitative variables, with p<.05 considered significant.

DETAILED DESCRIPTION:
The baseline interviews were conducted on the phone, on weekdays, during a mean time of 10 to 15minutes by a trained resident in psychiatry as the only interviewer. The interviewer didn't participate in patient's medical care nor in the follow-up interventions. The interviewer didn't look in patients file before conducted over the phone interviews and had only administrative information on the study subjects: first and last name, age, sex, phone number. The phone call interview wasn't considered as an intervention. Whenever the interviewer judged necessary that a patient needed more intensive treatment, the relevant referral to help was done.

ELIGIBILITY:
Inclusion Criteria:

* be male or female, be aged 18 or older, have a situation permitting follow-up contacts by phone.

Exclusion Criteria:

* be placed under supervision by the law such as guardianship and curatorship, be incarcerated and refusing to participate to the BCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The "Stay in contact" program concerns patients admitted to the PED for suicide attempt and who agree to benefit from this BCI
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
outpatients' experiences of the BCI "Stay in contact" | At the closure of the BCI Stay in contact, an average of 6 months after suicide attempt
  to assess the outpatients' experiences of the BCI "Stay in contact" using an hetero questionnaire completed over the phone by patients who benefited from the BCI.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Pichene, Principal Investigator — Psychiatric Emergency Departement, Central Hospital, Nancy, France; Fabienne Ligier, Principal Investigator — Psychiatric Emergency Departement, Central Hospital, Nancy, France; Sondos Abdalla, Principal Investigator — Psychiatric Emergency Departement, Central Hospital, Nancy, France
Locations (1):
- Central Hospital, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cedereke M, Monti K, Ojehagen A. Telephone contact with patients in the year after a suicide attempt: does it affect treatment attendance and outcome? A randomised controlled study. Eur Psychiatry. 2002 Apr;17(2):82-91. doi: 10.1016/s0924-9338(02)00632-6. PMID 11973116
- [Background] Hawton K, van Heeringen K. Suicide. Lancet. 2009 Apr 18;373(9672):1372-81. doi: 10.1016/S0140-6736(09)60372-X. PMID 19376453
- [Background] Hawton K, Saunders K, Topiwala A, Haw C. Psychiatric disorders in patients presenting to hospital following self-harm: a systematic review. J Affect Disord. 2013 Dec;151(3):821-30. doi: 10.1016/j.jad.2013.08.020. Epub 2013 Sep 7. PMID 24091302
- [Background] Gruat G, Cottencin O, Ducrocq F, Duhem S, Vaiva G. [Patient satisfaction regarding further telephone contact following attempted suicide]. Encephale. 2010 Jun;36 Suppl 2:D7-D13. doi: 10.1016/j.encep.2009.10.009. Epub 2009 Dec 1. French. PMID 20513463
- [Background] Milner A, Spittal MJ, Kapur N, Witt K, Pirkis J, Carter G. Mechanisms of brief contact interventions in clinical populations: a systematic review. BMC Psychiatry. 2016 Jun 8;16:194. doi: 10.1186/s12888-016-0896-4. PMID 27277833
- [Background] Castaigne E, Hardy P, Mouaffak F. [Follow-up interventions after suicide attempt. What tools, what effects and how to assess them?]. Encephale. 2017 Feb;43(1):75-80. doi: 10.1016/j.encep.2016.08.004. Epub 2016 Sep 28. French. PMID 27692348
- [Background] Kapur N, Cooper J, Bennewith O, Gunnell D, Hawton K. Postcards, green cards and telephone calls: therapeutic contact with individuals following self-harm. Br J Psychiatry. 2010 Jul;197(1):5-7. doi: 10.1192/bjp.bp.109.072496. PMID 20592425
- [Background] Pirkis J, Burgess P, Meadows G, Dunt D. Self-reported needs for care among persons who have suicidal ideation or who have attempted suicide. Psychiatr Serv. 2001 Mar;52(3):381-3. doi: 10.1176/appi.ps.52.3.381. PMID 11239110
- [Background] Burgess P, Pirkis J, Morton J, Croke E. Lessons from a comprehensive clinical audit of users of psychiatric services who committed suicide. Psychiatr Serv. 2000 Dec;51(12):1555-60. doi: 10.1176/appi.ps.51.12.1555. PMID 11097653
- [Background] Appleby L, Shaw J, Amos T, McDonnell R, Harris C, McCann K, Kiernan K, Davies S, Bickley H, Parsons R. Suicide within 12 months of contact with mental health services: national clinical survey. BMJ. 1999 May 8;318(7193):1235-9. doi: 10.1136/bmj.318.7193.1235. PMID 10231250
- [Background] Motto JA, Bostrom AG. A randomized controlled trial of postcrisis suicide prevention. Psychiatr Serv. 2001 Jun;52(6):828-33. doi: 10.1176/appi.ps.52.6.828. PMID 11376235
- [Background] Foster T, Gillespie K, McClelland R. Mental disorders and suicide in Northern Ireland. Br J Psychiatry. 1997 May;170:447-52. doi: 10.1192/bjp.170.5.447. PMID 9307695
- [Background] Hawton K et al. Attempted suicide : a practical Guide to its nature and management, 2nd ed. Oxford: Oxford University Press; 1987
- [Background] Kerkhof A al. Repetition of attempted suicide: results from the WHO/EU Multicentre Study on Parasuicide, repetition-prediction part. 7th European Symposium on Suicide and Suicidal Behaviour. Ghent: University Press; 1998
- [Background] Rygnestad T. [A 15-year follow-up study after deliberate self-poisoning]. Tidsskr Nor Laegeforen. 1997 Sep 10;117(21):3065-9. Norwegian. PMID 9381437
- [Background] Schmidtke A, Bille-Brahe U, DeLeo D, Kerkhof A, Bjerke T, Crepet P, Haring C, Hawton K, Lonnqvist J, Michel K, Pommereau X, Querejeta I, Phillipe I, Salander-Renberg E, Temesvary B, Wasserman D, Fricke S, Weinacker B, Sampaio-Faria JG. Attempted suicide in Europe: rates, trends and sociodemographic characteristics of suicide attempters during the period 1989-1992. Results of the WHO/EURO Multicentre Study on Parasuicide. Acta Psychiatr Scand. 1996 May;93(5):327-38. doi: 10.1111/j.1600-0447.1996.tb10656.x. PMID 8792901
- [Background] Gilbody S, House A, Owens D. The early repetition of deliberate self harm. J R Coll Physicians Lond. 1997 Mar-Apr;31(2):171-2. PMID 9131517
- [Background] Lönnqvist J et al.Suicide following the first suicide attempt: a five-year follow-up using a survival analysis. Psychiatr Fenn 1991;22:1719
- [Background] Van Heeringen K. The management of non-compliance with outpatient after-care in suicide attempters: a review. Ital J Suicidol 1992 ; 2 : 79-83
- [Result] Evans MO, Morgan HG, Hayward A, Gunnell DJ. Crisis telephone consultation for deliberate self-harm patients: effects on repetition. Br J Psychiatry. 1999 Jul;175:23-7. doi: 10.1192/bjp.175.1.23. PMID 10621764
- [Result] Vaiva G, Vaiva G, Ducrocq F, Meyer P, Mathieu D, Philippe A, Libersa C, Goudemand M. Effect of telephone contact on further suicide attempts in patients discharged from an emergency department: randomised controlled study. BMJ. 2006 May 27;332(7552):1241-5. doi: 10.1136/bmj.332.7552.1241. PMID 16735333
- [Result] Lebow JL. Client satisfaction with mental health treat- ment: Methodological considerations in assessment. Eval Rev 1983; 7:729-52
- [Result] Aoun S, Johnson L. A consumer's perspective of a suicide intervention programme. Aust N Z J Ment Health Nurs. 2001 Jun;10(2):97-104. doi: 10.1046/j.1440-0979.2001.00199.x. PMID 11421977
- [Result] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258